CLINICAL TRIAL: NCT00410371
Title: An Open-label, Randomised, Single-dose, Parallel-group Study to Evaluate the Pharmacokinetic Characteristics, Safety and Tolerability of up to Two Formulations (With Different Taste Masking Approaches) of an Orally Disintegrating Tablet (ODT) of Lamotrigine at 25mg and 200mg Versus the Immediate Release (IR) Lamotrigine in Healthy Subjects
Brief Title: Study to Compare Two Formulations of Lamotrigine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBI108614
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Mental Disorders
Keywords: tolerability; safety; Pharmacokinetic characteristics
MeSH Terms: conditions — Mental Disorders | interventions — Lamotrigine

ARMS (1):
- GI267119 (Experimental): 25 mg ODT tablet strength
  Interventions: Drug: Lamotrigine; Drug: GI267119

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine
Drug: GI267119 — 25 mg ODT

SUMMARY:
This study intends to compare the pharmacokinetic characteristics, safety and tolerability of two formulations of lamotrigine in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Body weight >50 kg (males) or >45 kg (females) and BMI within the range 19 to 30 kg/m2 inclusive.

Exclusion Criteria:

* Female subjects of childbearing potential will not be eligible to participate if they are unwilling or unable to use an appropriate method of contraception at least 30 days prior to the first study drug through 30 days.
* Female subject is pregnant (positive serum human chorionic gonadotrophin (hCG) test at Screening and pre-dose to the study) or lactating.
* Female subjects using hormonal contraceptive precautions including progesterone-coated intra-uterine device (IUD).
* Female subjects using hormonal replacement therapy.
* History of regular alcohol consumption
* Current smokers of 10 or more cigarettes per day

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2006-12-28 (Actual); Primary Completion 2007-01-25 (Actual); Study Completion 2007-01-25 (Actual)

PRIMARY OUTCOMES:
Lamotrigine AUC(0-inf) and Cmax | Time points when measures are taken : 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours

SECONDARY OUTCOMES:
tmax and t1/2, Adverse events, changes in biochemistry, haematology, urinalysis parameters, electrocardiogram parameters, blood pressure and heart rateTime points | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study LBI108614 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/LBI108614?search=study&search_terms=LBI108614#rs
- Available data/document: Informed Consent Form: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LBI108614 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register